CLINICAL TRIAL: NCT01632618
Title: Trunk Muscle Training and Neuromuscular Electrical Stimulation to Improve Function in Older Adults With Chronic Low Back Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Gregory Evan Hicks, Associate Professor, Physical Therapy, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 160167
Record Dates: First submitted 2012-06-28; First posted 2012-07-03 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trunk Muscle Training+NMES (Experimental): Progressive exercise program for the stabilizing muscles of the trunk, as well as neuromuscular electrical stimulation to the lumbar paraspinals
  Interventions: Behavioral: Trunk Muscle Training+NMES
- Passive control intervention (Active Comparator): Passive physical therapy interventions, including moist heat, ultrasound, massage and flexibility exercises
  Interventions: Behavioral: Passive control intervention

INTERVENTIONS:
Behavioral: Trunk Muscle Training+NMES — Progressive exercise program for the stabilizing muscles of the trunk, as well as neuromuscular electrical stimulation to the lumbar paraspinals
  Arms: Trunk Muscle Training+NMES
Behavioral: Passive control intervention — Passive physical therapy approach to low back pain
  Arms: Passive control intervention

SUMMARY:
Low back pain (LBP) is the most frequently reported musculoskeletal problem and third most frequently reported symptom of any kind in people over the age of 75. In fact, 17.3% of all visits to physicians for LBP involve individuals over 65. In older adults, LBP has been associated with a host of negative consequences, including decreased physical function, increased fall risk, increased mood disturbance and increased health care utilization. Surprisingly, little research has focused on LBP in people over 65. But, recent evidence demonstrates that LBP is associated with increased intramuscular fat infiltration in the abdominal and paraspinal muscles and that this altered muscle composition increases the risk of mobility-related functional decline in older adults. While trunk muscle training (TMT) has been used in younger LBP groups, it is unproven in elders and, alone may not be sufficient to substantially improve function and symptoms, given the compromised state of ages muscle. TMT augmented with neuromuscular electrical stimulation (NMES) known to improve strength and function beyond the capacity of volitional exercise alone, may provide greater improvements. Treatment of chronic LBP in older adults using an exercise intervention has been hypothesized as a way to prevent functional decline and frailty progression; however this hypothesis has yet to be experimentally confirmed. In this exploratory study, the investigators will test the hypothesis that TMT plus NMES will result in reduced disability and pain severity compared to usual care in elders with chronic LBP.

ELIGIBILITY:
Inclusion Criteria: 64 participants > age 65 will be recruited to participate. Participants will be included if they meet the following criteria:

- Low Back Pain for at least 3 months with pain of at least moderate intensity every day or almost every day that requires activity modification. This criterion is necessary to guarantee a subject population that has chronic pain that is not controlled with conventional therapy. At least moderate pain intensity (> 3 on a scale of 0-10) will be required to ensure our ability to detect treatment effects, and because pain of moderate intensity has been shown to be significant in the pain literature.11 The Pain thermometer has been shown to be reliable in older adults12, 13, will be used to screen pain intensity.

Exclusion Criteria:

* Exclusion Criteria: Subjects will be excluded from the study if any of the following exist:

  * Prominent component of radicular pain: CLBP with distal radiation below the knee
  * Known spinal pathology other than osteoarthritis: (e.g., a history of back surgery or recent trauma, spinal stenosis, vertebral compression fractures, ankylosing spondylitis, carcinoma metastatic to the spine) In these other cases, LBP may be of non-mechanical origin.
  * Non-ambulatory, or severely impaired mobility (i.e., require the use of a walker): Since measurement of physical performance in the proposed study includes gait velocity and standing balance, conditions other than LBP that could negatively impact these measures may confound our study results.
  * Folstein Mini-Mental State Examination score of < 24 will exclude subjects because of the uncertain reliability of their answers to the self-reported outcome measures.
  * Severe visual or hearing impairment: Since this study will involve questionnaires and telephone evaluations, severe visual and/or hearing impairments may interfere with data collection.
  * Red flags indicative of a serious disorder underlying the LBP: Red flags that would require specialized medical attention include fever, significant unintentional weight loss, a sudden recent change in the character or intensity of pain, trauma that preceded the onset of pain, or signs and symptoms of caudae equinae. These subjects will be promptly referred to their primary practitioners.
  * Significant pain in parts of the body other than the back or acute LBP: Since we will be specifically evaluating chronic LBP, we do not want to confound the outcome data with pain from other areas or with acute pain. Thus only subjects with LBP severity that is greater than pain severity elsewhere in the body will be included.
  * Acute or terminal illness: To insure weekly participation and a six month follow-up, subjects with an acute or terminal illness will be excluded from the study.
  * Presence of a pacemaker: Since electrical stimulation will be used in this study and the effects of that stimulation on pacemakers is unknown, we will be cautious and exclude subjects with this device.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go | 6 months
  timed performance test

SECONDARY OUTCOMES:
Gait speed | 6 months
Oswestry Low Back Pain Disability Questionnaire | 6 months
Global Rating of Functional Improvement | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregory E Hicks, PT, PhD, Principal Investigator — University of Delaware